CLINICAL TRIAL: NCT02515396
Title: A Randomised, Double-Blind, Placebo-Controlled, Two-Way Crossover Study in Healthy Smokers to Investigate the Effect of Inhaled Dosing With MMI-0100 on Airway Inflammation as Assessed in Induced Sputum After Challenge With Inhaled Lipopolysaccharide (LPS)
Brief Title: Phase 1a Study in Healthy Smokers to Investigate the Effect With MMI-0100 on Airway Inflammation in Induced Sputum After Challenge With Inhaled Lipopolysaccharide
Acronym: LPS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Moerae Matrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MMI-0100 RCT205
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Acute Inflammatory Response to Non-antigenic Stimulus
MeSH Terms: interventions — MMI-0100

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Experimental): MMI-0100 Inhaled, once daily x 5, followed by 3 week washout period, followed by Placebo Inhaled, once daily x 5
  Interventions: Drug: MMI-0100; Drug: Placebo
- Treatment Group B (Experimental): Placebo Inhaled, once daily x 5, followed by 3 week washout period, followed by MMI-0100 Inhaled, once daily x 5
  Interventions: Drug: MMI-0100; Drug: Placebo

INTERVENTIONS:
Drug: MMI-0100
Drug: Placebo

SUMMARY:
A Phase 1a, randomized, placebo controlled, two-way crossover study is to determine the effect of inhaled MMI-0100 compared to placebo following LPS challenge on inflammatory markers.

DETAILED DESCRIPTION:
The purpose of this Phase 1a, randomized, placebo controlled, two-way crossover study is to determine the effect of inhaled MMI-0100 compared to placebo on inflammatory markers following 5 days once daily (qd) dose of MMI-0100 or placebo administered by inhalation. On Day 5 of each treatment period, subjects will be challenged with inhaled LPS. Pharmacokinetics and biomarkers will be conducted at selected timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Written signed informed consent
* Comply with study procedures
* Body mass index (BMI) between 18 and 35 kg/m2 inclusive;minimum body weight of 50 kg
* Male subjects:

  1. Subjects with female partners of childbearing potential must agree to use a highly effective form of birth control, which entails the use of oral, injected or hormonal methods of contraception or intrauterine device/system by the female partner, in combination with a barrier method (e.g. condom, diaphragm, cervical cap with spermicide) during the study and for 3 months after discontinuation of treatment
  2. Subjects who are sterilised or have a female partner who is sterilised
  3. Subjects with a lifestyle that implies abstinence from sexual activity during the study and for 3 months after discontinuation of treatment
* Female subjects:

  1. Confirmed post-menopausal women (no periods for at least one year and follicle stimulating hormone (FSH) levels compliant with post-menopausal status according to reference values)
  2. Subjects agreeing to use highly effective form of birth control, which entails the use of oral, injected or implanted hormonal methods of contraception or intrauterine device/system in combination with a barrier method (e.g. condom, diaphragm, cervical cap with spermicide) during the study and for 3 months after discontinuation of treatment
  3. For females of childbearing potential: females must have a negative urine pregnancy test at screening and admission
* Normal physical examination, laboratory values, 12-lead electrocardiogram (ECG) and vital signs
* Be current smokers with defined smoking history of ≥10 pack years
* Ability to perform reproducible spirometry
* Demonstrate an FEV1 ≥80% of their predicted normal
* Demonstrate no evidence of airway obstruction
* Normal airway responsiveness to inhaled methacholine
* Have negative screens for serum hepatitis B surface antigen, Hepatitis C antigen and human immunodeficiency virus (HIV)
* Be able to produce a minimum of 0.1g sputum after induction with inhaled hypertonic saline at Visit 0

Exclusion Criteria:

* Subjects with an uncontrolled cardiovascular, respiratory, haematologic, immunologic, renal, neurologic, hepatic, endocrine disease, or any condition that might, in the judgment of the Investigator, place the subject at undue risk or potentially compromise the results or interpretation of the study
* Any clinically relevant abnormal value or physical finding that may interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part in the study
* Symptoms, signs or laboratory findings suggestive of an ongoing infective illness at the time of enrolment
* A history of respiratory disease including asthma
* Donation of more than 1200 mL of blood within 12 months of Visit 0 or, donation of blood in total >500 mL within 3 months prior to Visit 0
* Symptoms of any clinically significant illness within 2 weeks pior to Visit 0
* A significant history of alcohol abuse or consumption of more than 28 units (male) or 21 units (female) of alcohol per week
* A significant history of drug abuse (including benzodiazepines) or positive urine drugs of abuse test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 weeks
Cytokine Biomarkers | 6 weeks

SECONDARY OUTCOMES:
Neutrophil cell counts in sputum following LPS challenge | Within 1 day following challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinical Trials, The Heart Lung Centre, London, England, United Kingdom